CLINICAL TRIAL: NCT03016481
Title: Healing Through Education, Advocacy and Law (HEAL) in Response to Violence
Brief Title: Realizing Opportunities for Self-Supported Improvement (ROSSI)
Acronym: ROSE-SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Catherine Cerulli, Director of Susan B. Anthony Center for Women's Leadership and the Laboratory of Interpersonal Violence and Victimization, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IHS-1507-31543
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Domestic Violence; Depression; Quality of Life
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Community Health Worker -Personalized Support for Progress (Active Comparator): Patients will work with a Community Health Worker (CHW) to complete a prioritization tool and meet as needed over the course of the next 6 months to navigate services and overcome barriers. In addition, patients will receive referrals to other professionals based on their prioritization and meet with the CHW at the time and place of their choice.
  Interventions: Behavioral: Active Comparator: the Community Health Worker -Personalized Support for Progress
- Care as Usual- Social Worker (Active Comparator): Patients in the Care as Usual- Social Worker (CAU-SW) arm, will do intake with a social worker, who follows hospital procedures for intake and referrals, does a needs assessment, and offers safety planning in referral.
  Interventions: Behavioral: Care as Usual- Social Worker

INTERVENTIONS:
Behavioral: Active Comparator: the Community Health Worker -Personalized Support for Progress — Subjects will meet with their CHW to prioritize their needs detected by the Promote psychosocial screening and identify their preferences for intervention using a secure, online card sorting tool called Optimal Sort. The subject will explain her/his rationale for each decision to the CHW, allowing them both to begin to identify goals. The prioritization survey results provide subjects a personalized package of services that map onto the four main intervention options: legal help, problem solving therapy, medical consultation, or social services.
  Other Names: CHW-PSP
  Arms: the Community Health Worker -Personalized Support for Progress
Behavioral: Care as Usual- Social Worker — Based on their assessment and the subjects' needs, brief onsite interventions are provided and consist of empowerment focused advocacy, IPV education, community referrals, and safety planning. Participants determine follow-up. This will be a short-term interaction as routinely practiced across hospital settings.
  Other Names: CAU-SW
  Arms: Care as Usual- Social Worker

SUMMARY:
This is a 3-year comparative effectiveness study funded by the Patient Centered Outcomes Research Institute (PCORI) and will test an adapted priority-based patient navigation versus care as usual among 300 survivors of intimate partner violence (IPV) recruited from, and/or referred from, University of Rochester Medical Center providers. The goal is to improve patient safety, depression, and health function over the course of 12 months. In the Community Health Worker -Personalized Support for Progress (CHW-PSP) arm, created and tested in our first UR PCORI grant, in addition to meeting with a social worker, patients will work with a Community Health Worker (CHW) to complete a prioritization tool and meet as needed over the course of the next 6 months to navigate services and overcome barriers. In addition, patients will receive referrals to other professionals based on their prioritization and meet with the CHW at the time and place of their choice. Patients in the Care as Usual- Social Worker (CAU-SW) arm, will do intake with a social worker, who follows hospital procedures for intake and referrals, does a needs assessment, and offers safety planning in referral.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be English speaking URMC patients, who are 18 years of age or older, and/or the non-offending parent on a CPS report for a URMC pediatrics patient, and who have experienced an IPV or emotional abuse event within the past 3 months.

IPV is defined as endorsing any of the following items:

1. Slapped, kicked, pushed, choked, or punched?
2. Forced or coerced to have sex?
3. Threatened you with a knife or gun to scare or hurt you?
4. Made you feel afraid that you would be physically hurt?
5. Repeatedly used words, yelled, or screamed in a way that frightened you?
6. Threatened you, put you down, or made you feel rejected? Yes No Additional inclusion criteria include depression based on PHQ-9 score of >10.

Exclusion Criteria:

* Subjects are ineligible if they have active psychosis or alcohol or substance dependence based on 3 months threshold on the Mini-International Neuropsychiatric Interview (MINI).
* Additionally, patients who are unable to understand the consent form or study procedures, are imminently suicidal, or are currently working with a CHW will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Patient Safety | immediate post intervention (6 months)
  To assess whether CHW-PSP improves patient safety, as compared to CAU-SW Participants will complete the Conflict Tactics Scale-2 a modified from a 20-item self-report measure 10 assessing areas of negotiation, psychological aggression, physical assault, sexual coercion and injury. They will also complete the Danger Assessment, a 20-item measure to assess danger and lethality in a participant's experiences of violence and has documented reliability and validity. We will further assess safety with Steps for Safety instrument.The National Center for State Courts created the 18-item measure to document what safety steps a victim had taken post intervention. We will also receive Rochester Police Department (RPD) 911 call data, which is available to the public, and link the calls to our patients via address geomapping.
Depression | 9 months
  To assess whether CHW-PSP leads to improved depression and health function post-intervention (9 months). The PHQ-9 is a screen for major depressive disorder with good discriminant validity and sensitivity to change that has been validated in variety of settings.
Quality of Life | 12 months
  The effect of the Project Rose-SAFE intervention on the outcome of patient QoL will be mediated by increases in patient safety. The World Health Organization developed the WHOQOL-BREF to assess overall quality of life. It includes 4 summary scales: physical, psychological, social, and environment, plus a total score. The WHOQOL-BREF gives equal attention to the function and to a patient's assessment of the importance of that level of function, was designed to detect change over time, and is associated with change in depression.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cerulli, JD, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States